CLINICAL TRIAL: NCT03658863
Title: Comparison of Two Management Strategies, "Endoscopy First" and "Laparoscopic Cholecystectomy First", for Patients With Gallbladder Stones and Intermediate Risk for Choledocholithiasis
Brief Title: "Endoscopy First" or "Laparoscopic Cholecystectomy First" for Patients With Intermediate Risk of Choledocholithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Ausra Aleknaite, Investigator, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TLA02
Record Dates: First submitted 2018-08-13; First posted 2018-09-05 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Choledocholithiasis
Keywords: choledocholithiasis; endoscopic ultrasound; ERCP; intraoperative cholangiography; common bile duct stone; endoscopic retrograde cholangiopancreatography; gallstone disease; cholelithiasis; bile duct obstruction; laparoscopic cholecystectomy
MeSH Terms: conditions — Choledocholithiasis; Gallstones; Cholelithiasis; Cholestasis | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopy first (Active Comparator): Endoscopic ultrasound is used to evaluate bile ducts. If stones in extrahepatic bile ducts are seen ERCP and stone evacuation is performed during the same anaesthesia. Laparoscopic cholecystectomy is performed after endoscopic procedures in two days.
  Interventions: Procedure: endoscopic ultrasound; Procedure: ERCP; Device: Ultrasound endoscope
- Cholecystectomy first (Active Comparator): Laparoscopic cholecystectomy with intraoperative cholangiography is performed. If stones are found postoperative ERCP with stone evacuation is applied (during cholecystectomy if common bile duct is completely blocked or as soon as possible).
  Interventions: Procedure: intraoperative cholangiography; Procedure: ERCP

INTERVENTIONS:
Procedure: endoscopic ultrasound — Evaluation of bile ducts with endoscope with special ultrasonographic function
  Arms: Endoscopy first
Procedure: intraoperative cholangiography — evaluation of bile ducts by injecting radiocontrast media to cystic duct during laparoscopic cholecystectomy
  Arms: Cholecystectomy first
Procedure: ERCP — evaluation of bile ducts by injecting radiocontrast media to common bile duct via endoscope inserted to duodenum
  Other Names: endoscopic retrograde cholangiopancreatography
Device: Ultrasound endoscope — Endoscope with built-in ultrasound function
  Other Names: Endosonoscope
  Arms: Endoscopy first

SUMMARY:
The study compares two different methods to evaluate extrahepatic bile ducts for possible stones for patients with cholecystolithiasis and intermediate risk for choledocholithiasis when laparoscopic cholecystectomy is indicated.

Endosonoscopic evaluation of bile ducts and endoscopic retrograde cholangiography (ERCP) on demand are performed before laparoscopic cholecystectomy for one arm. Intraoperative cholangiography during laparoscopic cholecystectomy and postoperative ERCP on demand are administered in another arm.

DETAILED DESCRIPTION:
Use of ERCP as a diagnostic tool should be minimized as it carries considerable risk (5 to 10%) of post-procedural complications. It is noticed that adverse events occur more often to patients with low risk of choledocholithiasis. Therefore the best possible patient selection for ERCP procedure is needed.

At the Centre of Abdominal Surgery of Vilnius University Hospital Santaros klinikos an original prognostic index (Vilnius University Hospital index (VUHI)) is used for evaluation of risk of choledocholithiasis. It is calculated by formula VUHI = A/30 + 0.4×B, where A - total bilirubin concentration (µmol/l), B - common bile duct (CBD) diameter measured by ultrasound exam. A retrospective study evaluated its accuracy and determined threshold values for low, intermediate and high risk groups. The intermediate risk group (risk for choledocholithiasis 25-75%) would benefit from additional examination before ERCP. Endoscopic ultrasound (EUS) and intraoperative cholangiography are less invasive procedures with high accuracy identifying common bile duct stones. Main hypothesis of the trial is that intraoperative cholangiography with ERCP on demand can shorten the duration and costs of treatment and avoid diagnostic ERCPs.

ELIGIBILITY:
Inclusion Criteria:

* patients with cholecystolithiasis when laparoscopic cholecystectomy is indicated
* intermediate risk for choledocholithiasis (VUHI 2,6 - 6,9 and one of the predictors: dilated common bile duct, elevated total bilirubin or suspected stone in CBD on ultrasound)

Exclusion Criteria:

* pregnancy;
* acute cholangitis;
* biliary pancreatitis;
* acute cholecystitis, degree II-III by Tokyo guidelines 2013;
* anastomosis in upper gastrointestinal tract;
* other known cholestatic hepatopancreatobiliary disease;
* known or suspected hepatitis of another origin (viral, toxic, etc.);
* contraindications for general anaesthesia or surgery;
* IV-VI class of American Society of Anesthesiologists physical status classification;
* morbid obesity (body mass index > 40);
* patient's refusal to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Duration of treatment | up to one month
  duration from admission to hospital or decision to perform laparoscopic cholecystectomy to discharge in days

SECONDARY OUTCOMES:
Accuracy of different management strategies | 6 to 7 months
  Proportion of correctly diagnosed (true positive and true negative) cases in all sample
Technical success of interventions (IOC, EUS, ERCP) | up to one month
  For intraoperative cholangiography: successful cannulation and contrast media injection into CBD.
  For endoscopic sonoscopy: successful visualisation of CBD.
  For ERCP: successful cannulation and contrast media injection into CBD.
Adverse events of interventions | up to one month
  Bleeding, acute pancreatitis, perforation, allergic reactions
Costs of treatment | up to one month
  charges of diagnostic procedures, invasive procedures, surgery, antibacterial treatment if needed and hospital charges

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aleknaite A, Simutis G, Stanaitis J, Jucaitis T, Drungilas M, Valantinas J, Strupas K. Comparison of Endoscopy First and Laparoscopic Cholecystectomy First Strategies for Patients With Gallstone Disease and Intermediate Risk of Choledocholithiasis: Protocol for a Clinical Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 4;10(2):e18837. doi: 10.2196/18837. PMID 33538700